CLINICAL TRIAL: NCT00916968
Title: Comparison of Function and Fit of Standard Posterior Cruciate-Retaining High-Flexion and Gender-Specific Posterior Cruciate-Retaining High-Flexion Total Knee Prostheses A Prospective, Randomized Study
Brief Title: Comparison of Function and Fit of Standard and Gender-Specific CR High-Flex Total Knee Prostheses
Acronym: CR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ewha Womans University (Other)
Responsible Party: Young-Hoo, Kim M.D., Ewha Womans University Mokdong Hospital Joint Replacement Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2009-6-9
Record Dates: First submitted 2009-06-09; First posted 2009-06-10 (Estimated); Last update posted 2009-07-02 (Estimated); Status verified 2009-06

CONDITIONS: Osteoarthritis
Keywords: Gender specific; cruciate retaining; total knee arthroplasty; Bilateral Osteoarthritis of the knee joint
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard CR-Flex (Active Comparator)
  Interventions: Device: Standard CR-Flex total knee
- Gender specific CR-Flex (Experimental)
  Interventions: Device: Gender specific CR-Flex

INTERVENTIONS:
Device: Standard CR-Flex total knee — total knee implant used for joint replacement surgery of the knee
  Other Names: Zimmer, Nexgen CR-flex
  Arms: Standard CR-Flex
Device: Gender specific CR-Flex — TKA by Gender specific Nexgen CR-Flex
  Other Names: Gender Specific Nexgen CR-Flex implant
  Arms: Gender specific CR-Flex

SUMMARY:
The purpose of this prospective, randomized study was to compare functional outcome, radiographic results, range of motion, patients satisfaction, and fit of the femoral component in patients receiving either a standard posterior cruciate-retaining high-flexion (CR-flex) and gender-specific CR-flex total knee prostheses.

DETAILED DESCRIPTION:
The design features of the gender-specific knee prostheses have been claimed to improve fit and function of total knee arthroplasty in women. The purpose of this prospective, randomized study was to compare functional outcome, radiographic results, range of motion, patients satisfaction, and fit of the femoral component in patients receiving either a standard posterior cruciate-retaining high-flexion (CR-flex) and gender-specific CR-flex total knee prostheses.

ELIGIBILITY:
Inclusion Criteria:

* End stage osteoarthritis of the knee joint who require total knee arthroplasty with bilateral lesions.

Exclusion Criteria:

* Inflammatory arthritis
* Osteoarthritis effecting hip joint
* Traumatic arthritis
* Neurologic disorders affecting motor function of lower extremity
* foot and ankle disorders limiting ambulation of the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2007-02; Primary Completion 2007-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Knee Society Knee Score | 2 years

SECONDARY OUTCOMES:
Implant or bone overhang | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoowang Choi, MD, Principal Investigator — Ewha Womans University Mokdong Hospital
Locations (1):
- Ewha Womans University Mokdong Hospital, Seoul, South Korea